CLINICAL TRIAL: NCT06236906
Title: Digital-Physical Family Intervention in Primary Care for Families With Obesity in Both Children and Adults
Brief Title: Family Intervention for Treatment of Obesity With Digi-physical Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FamEv2024
Record Dates: First submitted 2023-12-20; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Childhood Obesity; mHealth; Personalized Medicine
Keywords: Obesity treatment; Digital support system
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Child and parent in digi-physical family treatment
  Interventions: Device: Device supported behavioural treatment

INTERVENTIONS:
Device: Device supported behavioural treatment — The method involves behavioral change supported by a digital support system, including daily home weighings, a clear weight curve in a mobile app, and communication with the treatment team through the same app.
  Other Names: Evira

SUMMARY:
Obesity in childhood is a global public health problem which continues to increase. It is associated with type 2 diabetes, high blood pressure, certain types of cancer, decreased psycho-social health and early mortality, among many other short- and long-term consequences. In many families where a child has obesity, at least one parent also has obesity or overweight with co-morbidity. In many cases, the care for children is more structured than for adults. Family treatment aimed at making lifestyle changes for the entire family, with those with obesity also restricting their calorie intake to normalize weight, has not been tested in Sweden and on a very limited scale internationally. International studies have shown that the more frequent the contact with healthcare, the better the results, regardless of the treatment method. However, frequent contacts are challenging to implement due to significant demands on both families and healthcare.

To address these challenges, the investigators aim to facilitate, improve, and optimize healthcare using a digital treatment support system involving daily home weighing and electronic communication between the clinic and families via a mobile application. The system is unique as it is based on real measurements, allowing both families and clinical staff to continuously monitor weight changes. This treatment involves fewer physical visits to the clinic but more frequent contact through the digital support system.

The goal is to evaluate whether a digital-physical family treatment conducted in primary care for families with at least one adult and one child with obesity leads to sustained weight loss with fewer visits, fewer missed appointments, resulting in more cost-effective care.

DETAILED DESCRIPTION:
The investigators have evaluated a digital support system for childhood obesity. The result shows twice as good results for the children who used the system compared to a control group treated with usual care despite a low frequency of physical clinical visits.

The method involves behavioral change supported by a digital support system, including daily home weighing, a clear weight curve in a mobile app, and communication with the treatment team through the same app. Working with the support system means that, as a caregiver, one follows a clear manual. The core idea is that families, using a partially Motivational Interviewing-based communication approach, find their own ways to reduce excess weight in accordance with what the mobile app indicates. The healthcare provider offers information as needed but refrains from providing specific advice. Instead, the provider supports how to manage the changes. Treatment focuses on the parental role, setting boundaries, collaboration, conflict resolution, and avoiding self-deception.

Over six months, 8-12 families will undergo Family Treatment within primary care. The goal is to evaluate the treatment's effectiveness based on experiences from both families and caregivers, using surveys and semi-structured interviews after three and six months.

ELIGIBILITY:
Inclusion Criteria:

* One or more children with obesity. Obesity defined based on the International Task Force criteria iso-BMI 30 and 35.
* At least one parent with obesity, i.e., BMI >30, or overweight with risk factors or comorbidity with a desire and willingness to lose weight.

Exclusion Criteria:

* Mental or physical illness in the child or parent that could seriously complicate the study's implementation.
* Serious language barriers preventing written communication in the digital support system.
* Separated parents where collaboration problems may complicate the study's implementation.
* Other reasons assessed to seriously complicate the study's implementation.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Families and practitioners experience of the treatment | Baseline, and at three and six months follow-up.
  Evaluate the experience from both families and practitioners regarding the treatment of the child and parent together with the support of the digital support system. Evira specific questionnaires.

SECONDARY OUTCOMES:
Families adherence to treatment | Trough study completion, an average of six months.
  Number of physical appointments, cancellations, and missed visits.
Families adherence in the use of the digital support system | Trough study completion, an average of six months.
  Frequency of Evira weighings, written and received messages
36-Item Short Form Survey (SF-36) for parents | Trough study completion, an average of six months.
  Questionnaires regarding quality of life. 36-Item Short Form Survey (SF-36) for parents. SF-36 cover eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. All items are scored so that a high score defines a more favorable health state.
Pediatric Quality of Life Inventory 4.0 for children (PedsQL) | Trough study completion, an average of six months.
  Pediatric Quality of Life Inventory 4.0 for children (PedsQL). PedsQL is a generic core scales instrument and contain 23-items in four scales, physical functioning, emotional functioning, social functioning, and school functioning. The higher scores indicate better health-related quality of life.
Participants', the children and parents psycho-social health during the family treatment | Trough study completion, an average of six months.
  Questionnaires regarding negative side effects such as the occurrence of eating disorders, anxiety, or depression (Evira specific questionnaires).
Change in BMI | At three and six months follow-up.
  Weight and height will be combined to report BMI in kg/m^2 for analyzing change in BMI Standard Deviation Score for the child and BMI for the parent.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
Using the evaluation from this study, we aim to optimize the family treatment method and finalize the application design based on user experiences for a larger randomized trial. as there are few individuals from a small place in Sweden, it will be difficult to keep the data anonymous.

REFERENCES:
- [Background] Johansson L, Hagman E, Danielsson P. A novel interactive mobile health support system for pediatric obesity treatment: a randomized controlled feasibility trial. BMC Pediatr. 2020 Sep 23;20(1):447. doi: 10.1186/s12887-020-02338-9. PMID 32967638
- [Background] Hagman E, Johansson L, Kollin C, Marcus E, Drangel A, Marcus L, Marcus C, Danielsson P. Effect of an interactive mobile health support system and daily weight measurements for pediatric obesity treatment, a 1-year pragmatical clinical trial. Int J Obes (Lond). 2022 Aug;46(8):1527-1533. doi: 10.1038/s41366-022-01146-8. Epub 2022 May 31. PMID 35641569
- See also: Evira homepage — http://www.evira.se/en/